CLINICAL TRIAL: NCT02163304
Title: Effects of Images Following Beverage Ingestion on Brain Activation
Acronym: Sweety
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, John Apolzan, Postdoctoral Fellow, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 2013-031
Record Dates: First submitted 2013-09-17; First posted 2014-06-13 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Sucrose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Artificial Sweetner (Active Comparator): Artificial Sweetener
  Interventions: Other: Artificial Sweetner
- Tasteless Solution (Placebo Comparator): 12 oz tasteless solution
  Interventions: Other: Tasteless Solution
- Sucrose (Active Comparator): 12 oz 75 g sucrose beverage
  Interventions: Other: Sucrose

INTERVENTIONS:
Other: Sucrose
  Arms: Sucrose
Other: Artificial Sweetner
  Arms: Artificial Sweetner
Other: Tasteless Solution
  Arms: Tasteless Solution

SUMMARY:
The primary purpose of this study is to quantify activation of regions of the brain associated with taste, appetite, and reward after viewing high sugar and high fat (HS/HF) images compared to control images following ingestion of (1) an artificially sweetened solution, (2) a sucrose solution, and (3) a tasteless control solution in normal weight vs. obese women. This is a repeated measures study design; hence, data are collected on three days corresponding to the three solutions. Body mass index (BMI) is a between subjects measure.

1. After consuming an artificially sweetened solution and a sucrose solution compared to a tasteless solution, viewing HS/HF food images vs. control images will result in higher activation of taste pathways (frontal operulum and anterior insula (FO/AI)) in the brain.
2. After consumption of a sucrose solution compared to an artificially sweetened solution and a tasteless solution, viewing HS/HF food images vs. control images will result in higher activation of regions of the brain associate with appetite (hypothalamus).
3. After consumption of a sucrose solution compared to an artificially sweetened solution and a tasteless solution, viewing HS/HF food images vs. control images will result in higher activation of regions of the brain associated with reward [amygdala, anterior cingulate cortex (ACC), Orbitalfrontal Cortex (OFC), and ventral tegmental area (VTA), striatum, insula] in obese but not normal weight women. After consuming an artificially sweetened solution compared to a tasteless solution, viewing HS/HF images vs. control images will result in no differences in activation of reward pathways of the brain.

DETAILED DESCRIPTION:
In this pilot study, we will use functional magnetic resonance imaging (fMRI) to determine the effects of high calorie visual food cues [i.e. images of foods that are high in both sugar and fat (HS/HF), such as ice cream] on activation of taste, appetite, and reward pathways in the brain following the separate ingestion of (1) an artificial sweetened solution (2) a sucrose solution and (3) a tasteless solution in obese individuals. Obesity rates are high among US adults with 33.8% of adults having a BMI of 30 or greater (1). The prevailing belief is that homeostatic systems are in place to monitor energy homeostasis. Sugar sweetened beverages appear to alter the homeostatic systems so that (1) metabolic feedback signals do not function correctly or as intended (2), as little or no dietary compensation is seen with energy from beverages (3), or (2) sweet and savory foods (sugar sweetened beverages) override the system (i.e. hedonics) (2). Epidemiological data suggest Americans are consuming 20-25% of their energy in beverage form which equates to ~430-535 kcal/day (3, 4). In most studies, sugar sweetened beverage intake has been shown to increase weight (5, 6). While limited data are available, a meta-analysis in humans demonstrates that the inclusion of aspartame compared to sugar reduces energy intake (7). A prospective study found that weight loss maintainers utilize artificial sweeteners more than normal weight individuals (8). This suggests artificial sweeteners may be a method to promote weight loss in obese individuals. Public policy on sugar sweetened beverages is starting to be reexamined, however, it is currently unknown what effect sugar sweetened beverage intake and artificial sweetened solutions have on (1) taste, appetite, and reward regions of the brain and (2) food cravings and related brain activation, among obese vs. normal weight individuals. The aim of this study is to provide important data on why obese individuals continue to consume sugar-sweetened beverages despite the associated negative health outcomes. We hypothesize that this consumption is due to sugar sweetened beverages, but not artificial sweeteners, activating reward pathways of the brain (hedonics).

Sucrose and artificial sweetners Previously it has been found that there is an altered hypothalamic response to glucose ingestion in obese humans (9). In obese humans, brain activation seems impaired; i.e., it was lower and delayed compared to lean subjects. This study lacked a functional contrast and had higher noise and less accuracy than current fMRI blood-oxygen-level-dependent (BOLD) technology and only the hypothalamus was analyzed (9). The current study and future studies from this pilot and feasibility work will further determine if dietary sugar responses are differentially regulated in obese individuals possibility contributing to the over consumption of sugar sweetened beverages in obese adults.

Frank et al. concluded that taste pathways are activated with sucralose and sucrose taste in younger normal weight women (10). Only sucrose recruited reward pathways but appetite pathways were not documented due to either lack of significance or examination (10). This study will confirm beverage ingestion opposed to tasting evokes a similar reward response and also examines appetite and reward pathways in obese individuals.

The effects of caloric vs. non caloric sweetener on taste activation were previously examined in normal weight men (11). During the non-caloric solution tasting, 2 caloric tastants were also consumed. These caloric tastants could invoke differential cephalic phase responses altering the results (12). Consumption of the artificial sweetener or the caloric solution increased activation of the insula, middle OFC, lateral OFC and amygdala. With the artificial sweetener, there was greater activation of the OFC (11). Next, the effects of sweet taste (2.4 mL) in younger male and female diet soda drinkers was examined (13). Water was utilized as the rinse and baseline for the comparison between diet and regular soda. In these persons, higher right orbitalfrontal cortex brain activation response in non-caloric compared to caloric solution was observed (13). These previous studies utilized only normal weight participants and taste to examine for the effects of artificial sweeteners on brain response. The current study examines obese individuals and solution ingestion to observe differences in brain activation. Overall there are differential brain responses to caloric vs. non-caloric sweetener in normal weight individuals thus previously authors suggested that more research needs to be performed as to the effectiveness of artificial sweeteners at decreasing energy intake.

Obesity Women were shown food picture cues of high energy foods. The high energy foods produced significantly greater activation in the brain reward regions in obese compared to normal weight control women (14). Differences between groups included ACC, VTA, nucleus accumbens (NAc), amygdala, ventral pallidum (Vent Pall), Caudate, and Putamen (14). Postmeal, obese individuals, but not normal weight individuals, increase activation of the putamen (part of striatum) and amygdala suggesting these regions may play a role in overeating (15) which is why these regions are incorporated into the current study hypothesis. These cross-sectional studies are important as previously Murdaugh et. al (16) found that obese individuals that were not successful at short term weight loss or longer term weight loss maintenance had greater activation of reward pathway brain regions. While speculative, artificial sweeteners may reduce cravings by not activating reward pathways especially in obese persons. This grant will help provide pilot data to further elucidate this important question.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 20-35 years old (inclusive)
* Weigh less than 350 lbs
* Weight stable (>±5 kg in the last 6 months).
* Body mass index (BMI) between 20-25 kg/m2 or 30-35 kg/m2.
* Willing to fast for 10 hours prior to examination.
* Right handed.

Exclusion Criteria:

* Diagnosis (by self report) of diabetes
* Diagnosis (by self report) of neurological condition
* Current or past alcohol or drug abuse problem.
* Smoking
* Have internal metal medical devices including cardiac pacemakers, aortic or cerebral aneurysm clips, artificial heart valves, ferromagnetic implants, shrapnel, wire sutures, joint replacements, bone or joint pins/rods/screws/clips, metal plates, metal fragments in your eye, or non-removable metal jewelry such as rings.
* Unable or unwilling to complete the imaging procedures for the duration of the MRI scan due to claustrophobia or other reason.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
fMRI | Visit 1,2,3
  fMRI will be performed using a General Electric Signa Excite HDxT 3.0T scanner (Milwaukee, WI) approximately 10 minutes post beverage ingestion. The field of view is 24-28 cm. The scanner is equipped with functional components from GE. Supplemental components include a projection system and eye imaging system from Avotec , Inc. An eight channel head coil will be utilized for all fMRI scans, and E-prime® software will be utilized for computerized experiment design, data collection, and analysis. Visual food and control cues will be presented in a mixed event block design with blocks of HS/HF and control images. Food cues consist of full-color pictures displaying foods within a category (HS/HF). One food item will be shown in each picture. Control cues consist of scrambled images that match the food cues in color intensity and frequency. Each block is 30s in length and 6 images are presented anywhere from 3-7seconds. Total task time will be ~30 minutes.

SECONDARY OUTCOMES:
VAS | Visit 1, 2, 3
  Visual Analog Scales (VAS). Paper VAS will be used to measure subjective ratings of hunger, satiety, fullness, prospective food consumption, and thirst during the present study. When completing the VAS, participants rate the intensity of subjective states or opinions on a line anchored from "not at all" to "extremely." The line is divided into 100 equal units. These VAS will be anchored from "strongly disagree" to "strongly agree." The VAS that measure appetite ratings will be completed at pre and post beverage preload and minute 60 (or immediately post scan) and 120 following the fMRI scan(s).

CONTACTS AND LOCATIONS:
Overall Officials: John W Apolzan, PhD, Principal Investigator — PBRC
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States